CLINICAL TRIAL: NCT04224922
Title: A Prospective, Belgian Multi-center, Single-arm, Phase II Study of Neoadjuvant Weekly Paclitaxel and Carboplatin Followed by Dose Dense Epirubicin and Cyclophosphamide in Stage II and III Triple Negative Breast Cancer
Brief Title: Phase II Study of Neoadjuvant Weekly Paclitaxel and Carboplatin Followed by Dose Dense Epirubicin and Cyclophosphamide in Stage II and III Triple Negative Breast Cancer
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: AZ-VUB (Other)
Collaborators: Universitaire Ziekenhuizen KU Leuven (Other); Universitair Ziekenhuis Brussel (Other)
Responsible Party: Principal Investigator, Dr Fontaine Christel, Principle Investigator, AZ-VUB
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: BSMO-2014-01
Record Dates: First submitted 2020-01-07; First posted 2020-01-13 (Actual); Last update posted 2020-01-18 (Actual); Status verified 2020-01

CONDITIONS: Breast Cancer
MeSH Terms: conditions — Breast Neoplasms | interventions — Paclitaxel; Carboplatin; Epirubicin; Cyclophosphamide

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- single-arm (Experimental): weekly paclitaxel at a dose of 80mg/m² in combination with weekly carboplatin (AUC=2), for 12 weeks, followed by 4 cycles of dose dense epirubicin at a dose of 90 mg/m² and cyclophosphamide at a dose of 600 mg/m² every 2 weeks (plus Long acting GCSF at day 2) administrated preoperatively in locally advanced operable stage II and III triple negative breast cancer
  Interventions: Drug: Paclitaxel; Drug: Carboplatinum; Drug: Epirubicin; Drug: Cyclophosphamide

INTERVENTIONS:
Drug: Paclitaxel
Drug: Carboplatinum
Drug: Epirubicin
Drug: Cyclophosphamide

SUMMARY:
This is a prospective Belgian, multi-center, open-label, single-arm phase II study of weekly paclitaxel at a dose of 80mg/m² in combination with weekly carboplatin (AUC=2), for 12 weeks, followed by 4 cycles of dose dense epirubicin at a dose of 90 mg/m² and cyclophosphamide at a dose of 600 mg/m² every 2 weeks (plus Long acting GCSF at day 2) administrated preoperatively in locally advanced operable stage II and III triple negative breast cancer to evaluate tumor response in the breast and the axilla.

ELIGIBILITY:
Inclusion Criteria:

* Stage II-III operable triple negative (ER and PR < 10%; Her2 IHC 0-1 or FISH <2.0) breast cancer in women age > 18. For patients aged 65 or older the G8 geriatric screening test should be > 14 (on a total of 17).
* Baseline mammography, US. MR of the breast on clinical indication.
* FNA of suspicious axillary lymph node is indicated
* Pre-treatment SN biopsy is indicated in clinical N0
* Measurable loco-regional disease
* Adequate bone marrow function, defined as

  * Absolute neutrophil count(ANC) >1500*109/L
  * Platelet count >100.000*109/L
* Adequate liver function defined as

  * Serum(total) bilirubin <1.5*upper limit of normal(ULN), unless the patient has documented Gilbert's Syndrome
  * AST and/or ALT <2.5*ULN
  * Alkaline phosphatase <2.5*ULN
* Normal cardiac function measured by ultrasound with a left ventricular function > 55%
* Creatinine clearance > 40 ml/min according to local laboratory standard (MDRD, CDK-epi, Cockroft-Gault, or other established formula to calculate renal function)

Exclusion Criteria:

* T4d breast tumor
* Bilateral breast cancer
* Other invasive cancer in the past except for a localized squamous cell cancer or basal cell of the skin or an in situ squamous cell cancer of the cervix.
* Pregnant or lactating patients

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 63 (Actual)
Dates: Start 2015-05 (Actual); Primary Completion 2016-07 (Actual); Study Completion 2017-05 (Actual)

PRIMARY OUTCOMES:
-The rate of pCR in the breast and axilla (ypT0/is, ypN0) | 20 weeks

SECONDARY OUTCOMES:
Evaluation of tumor infiltrating lymphocytes on the residual tumor | 20 weeks
  Histopathological analysis of the lymphocyte infiltrate is performed on hematoxylin and eosin- stained sections of the core biopsies and afterwords on the resection specimen after neoadjuvant chemotherapy. Ancillary techniques and immunohistochemistry have no additional value upon this date, and are not recommanded. The overall assessment has to be made for the whole tumor area, regardless of hot spots. All mononuclear cells including lymphocytes and plasma cells should be scored (granulocytes and other polymorphonuclear leukocytes are excluded). The quantitative assessment of other mononuclear cells such as dendritic cells and macrophages is currently not recommended. TILs should be reported for the intratumoral lymphocytes (as first proposed by Denkert in 2010). Stromal lymphocytes (Str-Ly) are defined as the percentage of tumor stroma area that contains a lymphocytic infiltrate without direct contact to tumor cells.
Number of participants with treatment-related adverse events as assessed by CTCAE v.4.03 | 20 weeks
Evaluation of the drug delivery | 20 weeks
  Patient compliance for paclitaxel and carboplatin and for epirubicin and cyclophosphamide will be assessed by the investigator and/or study personnel at each patient visit. To accurately determine the patient's drug exposure throughout the study, the following information must be reported on the Drug Administration Record CRF pages and in the source document.
  Planned dose administration, Actual total daily dose administrated, Regimen, Start and end date of drug administration, Dose change, Reason for dose change
Evaluation of clinical response rate (RECIST 1.1) by mammography and sonography in breast and axilla. | 20 weeks
Evaluation of breast-conserving surgery rate | 20 weeks
Evaluation of progression free survival | 20 weeks
Evaluation of overall survival | 20 weeks
Evaluation of percentage of patients with BRCA1 or BRCA2 in this population. | 20 weeks
genome analysis on tissue samples | 20 weeks
  Tumor tissue samples (FFPE) for genetic research will be obtained from consenting patients both at screening and at surgery.
  Genome analysis will be performed on (1) DNA extracted from EDTA blood (10ml) collected at the start of the treatment and (2) on DNA extracted from FFPE tumor tissue collected before the start of the neoadjuvant chemotherapy and after surgery.

CONTACTS AND LOCATIONS:
Overall Officials: Christel Fontaine, Dr., Principal Investigator — Universitair Ziekenhuis Brussel
Locations (18):
- Belgium (18):
  - Onze Lieve Vrouw Ziekenhuis, Aalst
  - Cliniques Sud Luxembourg, Arlon
  - Imelda Ziekenhuis, Bonheiden
  - AZ klina, Brasschaat
  - St Lucas, Bruges
  - Institut Jules Bordet, Brussels
  - Universitaire Ziekenhuis Antwerpen, Edegem
  - AZ Maria Middelares, Ghent
  - AZ St Lucas, Ghent
  - AZ Groeninge, Kortrijk
  - UZ Leuven, Leuven
  - CHR Citadelle, Liège
  - CHU Sart-Tilman, Liège
  - CMSE, Namur
  - Clinique st Pierre, Ottignies
  - CHWAPI, Tournai
  - CHR Verviers, Verviers
  - CHU Mont-Godinne, Yvoir